CLINICAL TRIAL: NCT02383498
Title: A Randomized, Double-Blind, Phase 2 Trial of GI-6301 (Yeast-Brachyury Vaccine) Versus Placebo in Combination With Standard of Care Definitive Radiotherapy in Locally Advanced, Unresectable, Chordoma
Brief Title: QUILT-3.011 Phase 2 Yeast-Brachyury Vaccine Chordoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QUILT-3.011
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2019-10

CONDITIONS: Chordoma
Keywords: Overall Response Rate; Immune Activation; Tumor Infiltrating Lymphocytes; T Cell Response; Cross-Over
MeSH Terms: conditions — Chordoma | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GI-6301 Vaccine (Experimental): Radiation + GI-6301 Vaccine + Actigraph
  Interventions: Biological: GI-6301 Vaccine (Yeast- Brachyury); Radiation: Radiotherapy; Device: wGT3X-BT Actigraph
- Placebo (Placebo Comparator): Radiation + Placebo + Actigraph
  Interventions: Other: Placebo; Radiation: Radiotherapy; Device: wGT3X-BT Actigraph

INTERVENTIONS:
Other: Placebo — Placebo will consist of USP-grade or equivalent 0.9% Sodium Chloride for Injection. Doses of placebo will be drawn into labeled syringes by an independent, unblinded pharmacist or designee.
  Arms: Placebo
Biological: GI-6301 Vaccine (Yeast- Brachyury) — GI-6301 Vaccine is a heat-killed, recombinant yeast-based vaccine engineered to express the transcription factor, Brachyury. The Brachyury gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wildtype yeast) to produce the final recombinant vaccine product.
  Arms: GI-6301 Vaccine
Radiation: Radiotherapy — Standard of care
Device: wGT3X-BT Actigraph — wGT3X-BT is small, non-invasive, portable watch accelerometer worn on the subject's wrist for Cycle 1 through Cycle 9

SUMMARY:
This is a phase 2 clinical trial to determine whether the yeast-brachyury vaccine GI-6301 improves the effectiveness of radiation for patients with localized chordoma. Chordoma patients with inoperable or residual tumor who do not have metastases and are planning to be treated with definitive (>70Gy) radiation were enrolled. Patients were randomized to receive radiation plus the vaccine or radiation plus a blinded placebo. The study compared the outcomes of patients treated with radiation with and without the vaccine to determine whether the vaccine can increase the chances of shrinking the tumor and/or preventing further tumor growth.

DETAILED DESCRIPTION:
Chordoma is a rare disease, affecting about 3,000 people in the United States. There have been indications of clinical benefit in patients with chordoma enrolled on the phase I trial of GI-6301.

PRIMARY OBJECTIVE: To determine if there is a difference in overall response rate (ORR) defined as complete response (CR) or partial response (PR) by RECIST 1.1 after up to 24 months among patients with Chordoma who are treated with radiation plus placebo vs. radiation plus vaccine.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet the following criteria for participation:

1. Diagnosis: Patients must have histologically confirmed chordoma by the Laboratory of Pathology, NCI, which is localized (no evidence of metastatic disease), unresectable and they must have planned radiation therapy, to at least one targeted lesion with evidence of growth prior to enrollment. The tentative radiation plan at enrollment must be in compliance with the required radiation doses. This can be given in standard or hypofractionated dosing with any technique deemed most appropriate by the treating radiation oncologist if other requirements are not met.
2. Patients must have disease that is measurable by RECIST version 1.1.
3. Fresh or archived tumor specimen must be available for correlative studies.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at study entry (Karnofsky greater than or equal to 70)
5. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of GI-6301 (Yeast Brachyury vaccine) in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
6. Prior Therapy: Patients must have fully recovered from prior surgery before enrollment. Prior radiation therapy is allowed provided the radiation field can safely irridated in the opinion of the treating radiation oncologist.
7. Patients must have normal organ and marrow function as defined below:

   * Serum creatinine less than or equal to 1.5 X upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 60 mL/min.
   * ALT and AST less than or equal to 3 X the upper limits of normal.
   * Total bilirubin less than or equal to 1.5 X upper limit of normal OR in patients with Gilbert s syndrome, a total bilirubin less than or equal to 3.0.
   * Hematological eligibility parameters (within16 days of starting therapy):

   Granulocyte count greater than or equal to 1,500/mm3

   Platelet count greater than or equal to 100,000/mm3
8. Men and women of child-bearing potential must agree to use effective birth control or abstinence during and for a period of 4 months after the last vaccination therapy.
9. Patients must not have a history of yeast allergy. If patient has a questionable history of allergy to yeast, a yeast skin test can be performed. Patients would be eligible if skin test is negative.
10. Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with any of the following will not be eligible for participation in this study:

1. Patients should have no evidence of immune dysfunction as listed below.

* Human immunodeficiency virus (HIV) positivity due to the potential for decreased immune response to the vaccine.
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. However, patients with vitiligo, diabetes mellitus, and Hashimoto thyroiditis on appropriate replacement therapy may be enrolled.
* History of allergy or untoward reaction to yeast-based products (any hypersensitivity to yeast-based products will be excluded).
* Pregnant or breast-feeding women, due to the unknown effects of the Yeast-brachyury vaccine on the fetus or infant.
* Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.
* Chronic hepatitis infection, including B and C, because potential immune impairment caused by these disorders may diminish the effectiveness of this immunologic therapy.
* Any significant disease that, in the opinion of the investigator, may impair the patient s tolerance of study treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Patients may not be on systemic steroids within 4 weeks of enrolling on study with the exception of physiologic replacement doses (for instance in the case of adrenal insufficiency) or steroid premedication for baseline MRI and/or CT in the case of subjects with known contrast dye allergies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0118.html
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8100546/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Radiation + GI-6301 Placebo + Actigraph
  GI-6301 Placebo: GI-6301 Placebo will consist of USP-grade or equivalent 0.9% Sodium Chloride for Injection. Doses of GI-6301 placebo will be drawn into labeled syringes by an independent, unblinded pharmacist or designee.
  Radiotherapy: Standard of care
  wGT3X-BT Actigraph: wGT3X-BT is small, non-invasive, portable watch accelerometer worn on the subject's wrist for Cycle 1 through Cycle 9
Period: Overall Study
Arm/Group | GI-6301 Vaccine | Placebo
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vaccine: Radiation + GI-6301 Vaccine + Actigraph
  GI-6301 Vaccine (Yeast- Brachyury): GI-6301 Vaccine is a heat-killed, recombinant yeast-based vaccine engineered to express the transcription factor, Brachyury. The Brachyury gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wildtype yeast) to produce the final recombinant vaccine product.
  Radiotherapy: Standard of care
  wGT3X-BT Actigraph: wGT3X-BT is small, non-invasive, portable watch accelerometer worn on the subject's wrist for Cycle 1 through Cycle 9
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 75] | 61 [48 to 76] | 61 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Subjects with Locally Advanced, Unresectable, Chordoma [Count of Participants; unit: Participants] | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Difference in overall response rate among patients with Chordoma who are treated with radiation plus placebo vs. radiation plus vaccine.
  Overall response rate (ORR) defined as complete response (CR) or partial response (PR) by RECIST 1.1 in the irradiated tumor site after up to 24 months among patients with Chordoma who are treated with radiation plus vaccine vs. radiation plus placebo
  Complete response (CR; disappearance of all target lesions and no new lesions) or partial response (PR; >=30% decrease in the sum of the greatest diameter).
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | GI-6301 Vaccine | Placebo
Number analyzed (Participants) | 11 | 13
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were to be reported within 30 days of last dose of administration, up to 219 weeks. For serious adverse events that occurred more than 30 days after the last administration of investigational agent/intervention, only reported those that had an attribution of at least possibly related to the agent/intervention.
Arm/Group | GI-6301 Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 5/11 | 1/13
Other Adverse Events (participants affected / at risk) | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GI-6301 Vaccine (N=11) | Placebo (N=13)
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Infections and infestations) | 1 | 0
Hyponatremia (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GI-6301 Vaccine (N=11) | Placebo (N=13)
Lymphocyte count decreased (Investigations) | 9 | 11
White blood cell decreased (Investigations) | 4 | 5
Alanine aminotransferase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 2
Creatinine increased (Investigations) | 2 | 3
Weight loss (Investigations) | 4 | 1
Alkaline phosphatase increased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 1
Weight gain (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Injection site reaction (General disorders) | 10 | 6
Fatigue (General disorders) | 6 | 8
Pain (General disorders) | 4 | 6
Flu like symptoms (General disorders) | 1 | 4
Edema limbs (General disorders) | 1 | 3
Gait disturbance (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 2
Fever (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Neck edema (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 5 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 3
Burn (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 6
Headache (Nervous system disorders) | 3 | 5
Paresthesia (Nervous system disorders) | 2 | 5
Dizziness (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 2
Stroke (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoglossal nerve disorder (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 2 | 2
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hot flashes (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 2
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 2
Floaters (Eye disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02383498/Prot_SAP_000.pdf